CLINICAL TRIAL: NCT03225625
Title: Stem Cell Spinal Cord Injury Exoskeleton and Virtual Reality Treatment Study
Acronym: SciExVR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MD Stem Cells (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SciExVR
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Spinal Cord Compression; Spinal Cord Ischemia; Spinal Cord Diseases; Spinal Paralysis; Paraplegia; Paraplegia, Spinal; Paraplegia/Paraparesis; Paraplegia; Traumatic; SCI - Spinal Cord Injury
Keywords: spinal cord injury; spinal cord compression; spinal cord ischemia; spinal cord diseases; spinal paralysis; paraplegia; paraparesis; SCI
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Compression; Spinal Cord Ischemia; Spinal Cord Diseases; Paraplegia; Paraparesis | interventions — DMAC2L protein, human

STUDY DESIGN:
Intervention Model Description: There will be 3 Arms:
  Arm 1: BMSC Paraspinal, IV, Intranasal . Arm 2: BMSC Paraspinal,IV,Intranasal + exoskeleton or equivalent . Arm 3: BMSC Paraspinal, IV, Intranasal + virtual reality or equivalent .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paraspinal (Experimental): Bilateral paraspinal injection of bone marrow derived stem cells (BMSC) at spinal cord injury level, superior to injury level and inferior to injury level. Following paraspinal injection remaining BMSC provided intravenous and intranasal.
  Interventions: Procedure: Paraspinal
- Paraspinal EX (Experimental): Bilateral paraspinal injection of bone marrow derived stem cells (BMSC) at spinal cord injury level, superior to injury level and inferior to injury level. Following paraspinal injection remaining BMSC provided intravenous and intranasal.
  Exoskeleton or equivalent stimulation following this treatment.
  Interventions: Procedure: Paraspinal; Procedure: Paraspinal EX
- Paraspinal VR (Experimental): Bilateral paraspinal injection of bone marrow derived stem cells (BMSC) at spinal cord injury level, superior to injury level and inferior to injury level. Following paraspinal injection remaining BMSC provided intravenous and intranasal.
  Virtual Reality or equivalent visualization following this treatment.
  Interventions: Procedure: Paraspinal; Procedure: Paraspinal VR

INTERVENTIONS:
Procedure: Paraspinal — BMSC provided by paraspinal injection, intravenous and intranasal
  Other Names: Arm 1
Procedure: Paraspinal EX — BMSC provided by paraspinal injections, intravenous and intranasal followed by exoskeleton or equivalent stimulation
  Other Names: Arm 2
  Arms: Paraspinal EX
Procedure: Paraspinal VR — BMSC provided by paraspinal injections, intravenous and intranasal followed by virtual reality or equivalent visualization
  Other Names: Arm 3
  Arms: Paraspinal VR

SUMMARY:
The SciExVR study will evaluate the potential benefit of autologous bone marrow derived stem cells (BMSC) in the treatment of spinal cord injury with evidence of impaired motor or sensory function. The treatment consists of bilateral paraspinal injections of the BMSC at the level of the injury as well as superior and inferior to that spinal segment followed by an intravenous injection and intranasal placement. Patients undergoing BMSC treatment may also be assigned to use of exoskeletal movement (or equivalent) or virtual reality visualization (or equivalent) to augment upper motor neuron firing and/or receptivity of the sensory neurons. http://mdstemcells.com/sciexvr/

DETAILED DESCRIPTION:
The Stem Cell Spinal Cord Injury Exoskeleton and Virtual Reality (SciExVR) study is based on the progress that researchers have made treating spinal cord injury (SCI) with bone marrow derived stem cells (BMSC). While major improvements have remained elusive with other approaches, modest benefits have been achieved.

The use of subarachnoid BMSC provided via intrathecal injection has resulted in improvements for certain sensory and bladder functions. Exoskeleton treatment has shown certain benefits in sensory, bowel and bladder function.

Intravenous (IV) BMSC have benefited stroke and other central nervous system damage. In the sponsor's concomitant Neurologic Stem Cell Treatment (NEST) study for general neurologic disease, benefit has been shown by combining IV with intranasal BMSC.

The SciExVR study uses paraspinal injections- meaning the BMSC are placed adjacent to the spinal nerves which enter the spinal canal through the intervertebral foramen of the vertebral bodies. The BMSC will be placed at the level of the injury on both sides of the spine as well as approximately two segments above and two segments below. The investigators believe this will allow entry into the spinal tissue at the injury site as well as to the injured upper motor neuron pathways; lower motor neurons which may be injured; sensory pathways; dorsal root ganglia at and below the site and autonomic ganglia. Placement in the paraspinal tissue may extend the time that BMSC have to proliferate at, above and below the vicinity of the spinal cord injury and interact with damaged cells in the spinal cord, spinal roots, spinal nerves and paravertebral ganglion. Potential benefits of these interactions include BMSC mitochondrial transfer to target cells, secretion of mRNA increasing target cell activity, secretion of nerve growth factor and other neurotrophic factors beneficial to nerve regrowth. Increased proliferation and contact time may increase neuronal transdifferentiation of BMSC to neurons and/or neuroglia. Following paraspinal injections the patient receives the remaining BMSC intravenously (IV) and also topically intranasally. BMSC given IV may enter the central nervous system through the paraventricular organs in the brain to potentially reach the ascending and descending pathways, thalamus, sensory cortex, motor cortex and circulate through the cerebral spinal fluid (CSF). Intranasal provides access through the axons of the Trigeminal (V) cranial nerves and entry into the brain at the level of the pons with similar opportunity to move through the tissues.

BMSC are separated from bone marrow obtained from the posterior iliac crest with a single aspiration on each side. The procedure is performed under general or MAC anesthesia at the fully licensed surgical center so there is no discomfort in performing the procedure. The BMSC are separated from the aspirate using an FDA cleared class II device.

After BMSC treatment patients who are in Arm 1 simply follow up with their own neurologists at 1,3,6 and 12 months.

Those in Arm 2 require similar follow up and pursue treatment at centers that can provide exoskeletal stimulation or physical therapy equivalent. Exoskeleton devices move the limbs of the patient to provide stimulation to the muscles in a self directed fashion but similar to physical therapy that is often performed for SCI. The investigators believe that Arm 2 may provide stimulation of the upper and lower motor neurons and sensory receptors such as exteroceptors and proprioceptors which may, in the presence of BMSC, assist in regeneration or reactivation of the spinal cord pathways.

Patients in Arm 3 require similar follow up and may use Virtual Reality headsets or equivalent to increase visualization of movement of the lower extremities and/or sensory feedback. This may also help stimulate the upper and lower motor neurons and sensory receptors.

ELIGIBILITY:
Inclusion Criteria:

* Have documented functional damage to the spinal cord unlikely to improve with present standard of care.
* If under current medical therapy (pharmacologic or surgical treatment) for the condition be considered stable on that treatment and unlikely to have reversal of the associated spinal cord damage as a result of the ongoing pharmacologic or surgical treatment.
* In the estimation of Dr. Weiss and Dr. Silberfarb have the potential for improvement with BMSC treatment and be at minimal risk of any potential harm from the procedure.
* Be over the age of 18 and capable of providing informed consent.
* Be medically stable and able to be medically cleared by their primary care physician or a licensed primary care practitioner for the procedure. Medical clearance means that in the estimation of the primary care practitioner, the patient can reasonably be expected to undergo the procedure without significant medical risk to health.

Exclusion Criteria:

* All patients must be capable of an adequate neurologic examination and evaluation to document the pathology. This will include the ability to cooperate with the exam.
* Patients must be capable and willing to undergo follow up neurologic exams as outlined in the protocol.
* Patients must be capable of providing informed consent.
* In the estimation of Dr. Weiss and Dr. Silberfarb the BMSC collection and treatment will not present a significant risk of harm to the patient's general health or to their neurologic function. .
* Patients who are not medically stable or who may be at significant risk to their health undergoing the procedure will not be eligible.
* Women of childbearing age must not be pregnant at the time of treatment and should refrain from becoming pregnant for 3 months post treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) Impairment Scale (AIS) | Pre-procedure, 1,3,6 and 12 months post-procedure
  AIS is based on the Frankel scale which is used to classify the degree or completeness of spinal cord injury (SCI) by assessing motor and sensory function. Patients will have AIS assessment prior to procedure and post-procedure for comparison and identification of any improvements in motor or sensory function.

SECONDARY OUTCOMES:
Autonomic Nervous System (ANS) Function | 1,3,6 and 12 months post-procedure
  The autonomic nervous system (ANS) through the sympathetic and parasympathetic divisions is responsible for many functions of the body including bladder and bowel control and sweating. Patients will self-report changes in ANS function and their abilities to perform ANS functions following the procedure.
General Well-Being | 1,3,6,12 months post-procedure
  General Well-Being is a term that may encompass mood, sense of well-being, family relationships, ability to do daily tasks and other practical or emotional practices that vary from person to person. Patients will self-report changes in their Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Steven Levy, MD, Study Chair — MD Stem Cells; Jeffrey Weiss, MD, Principal Investigator — Coral Springs; Steven Silberfarb, DO, Principal Investigator — Florida Orthopaedics and Spine Center
Locations (1):
- MD Stem Cells, Coral Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: No